CLINICAL TRIAL: NCT02840695
Title: Effect of Biological Disease Modifying Anti Rheumatic Drug (bDMARD) Treatment on Spinal Fracture Incidence in Patients With Ankylosing Spondylitis (AS)
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: bDMARD AS Spinal Fractures
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Ankylosing Spondylitis; Spinal Fractures
MeSH Terms: conditions — Spondylitis, Ankylosing; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AS patients: Patients registered in the Swedish Patient Registry with active AS treated with or without biological DMARD according to the Swedish Prescribed Drugs Registry, with or without spinal fractures
  Interventions: Drug: bDMARD treatment

INTERVENTIONS:
Drug: bDMARD treatment — Treatment with bDMARD includes registered ATC-codes: L04AA and L04AB.
  Other Names: Biological Disease Modifying Drug treatment

SUMMARY:
Ankylosing spondylitis (AS) is a rheumatoid disease affecting all segments of the axial skeleton, leading to the complete fusion of all spinal segments - the bamboo-spine. During the last decade biological disease modifying anti-rheumatic drugs (bDMARD) have been successfully introduced to reduce the disease activity. It is unclear whether bDMARD treatment had an effect on spinal fracture risk related to AS. This national registry study will investigate the effect of bDMARD treatment on spinal fracture risk in a national cohort of patients with AS.

ELIGIBILITY:
Inclusion Criteria:

* age 30-60 years
* registered diagnosis of ankylosing spondylitis

Exclusion Criteria:

* age <30 or >60 years

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with AS as registered in the Swedish Patient Registry with ICD-9-code 720 or ICD-10 code M45.9.
Sampling Method: Non-Probability Sample
Enrollment: 9858 (Actual)
Dates: Start 2005-01; Primary Completion 2015-12 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Spinal fracture | 10 years
  Censored data with occurrence of spinal fracture within 10 years observation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robinson Y, Olerud C, Willander J. Do biological disease-modifying antirheumatic drugs reduce the spinal fracture risk related to ankylosing spondylitis? A longitudinal multiregistry matched cohort study. BMJ Open. 2017 Dec 28;7(12):e016548. doi: 10.1136/bmjopen-2017-016548. PMID 29288176
- [Derived] Badar F, Mahmood S. Epidemiology of cancers in Lahore, Pakistan, among children, adolescents and adults, 2010-2012: a cross-sectional study part 2. BMJ Open. 2017 Dec 21;7(12):e016559. doi: 10.1136/bmjopen-2017-016559. PMID 29273649